CLINICAL TRIAL: NCT00397839
Title: A Parallel, Placebo-controlled, Randomized (2:1) Double-blind Study of One Year Duration to Assess the Effect of Oral Ibandronate 150 mg Given Once-monthly Versus Placebo on LS BMD in Men With Osteoporosis
Brief Title: The Effect Of Oral Ibandronate In Male Osteoporosis
Acronym: STRONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BON105960
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-11

CONDITIONS: Male Osteoporosis
Keywords: male osteoporosis; osteoporosis; bisphonates; bone
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Ibandronate (Experimental)
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Ibandronate orally (tablet) at a dose of 150 mg once per month
  Arms: Ibandronate
Drug: placebo — Placebo orally (tablet) at a dose of 150 mg once per month
  Arms: Placebo

SUMMARY:
Male osteoporosis is a common and important clinical problem, associated with significant morbidity, mortality and societal expense. Approximately 10% of men =65 years of age are osteoporotic. The proposed study will evaluate efficacy and safety of oral ibandronate given 150 mg once-monthly for 12 months versus placebo in men with primary osteoporosis. Less frequent, once monthly, dosing is expected to improve patient's treatment adherence compared to a weekly dosing regimen.

ELIGIBILITY:
Inclusion criteria:

* Ambulatory men at least 30 years old at screening, who are diagnosed with primary, idiopathic or hypogonadal osteoporosis according to the following criteria: Femoral neck (FN) BMD T-score < -2.0 and LS BMD T-score < -1.0 OR LS BMD T-score < -2.0 and FN BMD T-score < -1.0 and BMD T-score > 4.0 at any site
* Subjects who, in the opinion of the investigator, are willing and able to comply with the protocol requirements
* Subjects who have signed an informed consent

Exclusion criteria:

* Significant medical conditions or laboratory abnormalities, which in the opinion of the investigator may preclude the patient's ability to complete the study
* Malignant disease diagnosed within the previous 5 years (except resected basal cell cancer)
* Disease/disorder known to influence bone metabolism or cause of secondary osteoporosis e.g., chronic gastrointestinal or liver disease, renal disease, chronic alcoholism, malabsorption syndrome
* Hypersensitivity to any component of ibandronate
* Inability to stand or sit in an upright position for at least 60 minutes
* Inability to swallow a tablet without breaking it
* Vitamin D deficiency (serum 25-OH vitamin D <20ng/mL (equivalent to 50nmol/L) at screening
* Any prevalent osteoporotic vertebral fracture identified by total spine x-ray (Total spine x-ray consists of lateral and PA films of the thoracic & lumbar spine)
* Subjects who are receiving testosterone supplementation for < 2 years (if applicable) (Patients who are identified with clinical signs of hypogonadism at screening and are started on testosterone supplementation will be excluded from participation.)
* Contraindications to calcium or vitamin D therapy
* Administration of any investigational drug within 30 days preceding the first dose of the study drug
* Previous treatment with an oral bisphosphonate within the last six months, OR more than one month of cumulative treatment within the last year, OR more than three months of cumulative treatment within the last two years AND/OR treatment with intravenous bisphosphonate within one year.
* Treatment with PTH or similar anabolic agent for osteoporosis within the last two years
* Treatment with other drugs affecting bone metabolism within the last six months prior to Screening including:

  * Chronic systemic glucocorticoid treatment except for topical treatment at a frequency of up to twice per week
  * Calcineurin inhibitors [e.g., cyclosporine, tacrolimus] or methotrexate
  * Testosterone therapy (unless stabilized on medications > 2 years)
  * Calcitonin
  * Fluoride (dose greater than 10mg/day) or strontium for osteoporosis within the last 12 months, or past treatment for more than a total of 2 years
  * Selective estrogen receptor modulators (SERMS) such as raloxifene, toremifene, tamoxifen, arzoxifene and lasofoxifene
  * Anabolic steroids and other androgens, such as dehydroepiandrosterone (DHEA) or its sulphated form (DHEAs)
  * Active vitamin D analogs/metabolites such as1,25-dihydroxy vitamin D (calcitriol) or 1-alpha-hydroxy vitamin D3 (1 - alpha hydroxycholecalciferol)
  * Gonadotropin releasing antagonists (lupron)
* ALT > twice upper limit of normal range of central laboratory
* Hypercalcemia or uncorrected hypocalcemia: Serum total Ca 2+ > 10.5mg/dl or < 8.0 mg/dL (equivalent to 2.6 and 2.0 mmol/L)
* GFR < 30 ml/min as determined by estimated creatinine clearance (CLcr) calculated by the Cockcroft-Gault equation:

CLcr = (140-age) * ABW X 0.85 72*Scr where : CLcr - estimated creatinine clearance Age - in years ABW - actual body weight at screening (kg) Scr - serum creatinine at screening (mg/dL)

* History of major upper GI disease defined by:

  * Significant upper GI bleeding within the last year requiring hospitalization or transfusion
  * Recurrent peptic ulcer disease documented by radiographic or endoscopic means
  * Dyspepsia or gastroesophageal reflux that is uncontrolled by medication
  * Abnormalities of the esophagus that delay esophageal emptying, such as stricture, achalasia, or dysmotility
  * Active gastric/duodenal ulcers
  * Dyspepsia controlled by daily medication OR prior history of non-recurrent peptic ulcer disease are not considered exclusionary
* WBC < 2500/µL
* Serum albumin < 3.0g/dL
* History of hyperthyroidism, hyperparathyroidism or osteomalacia within one year of study entry
* Fewer than three (3) vertebrae in the range L1-L4 evaluable by DXA. Conditions which interfere with the BMD measurement include prevalent fracture, sequelae of orthopedic procedures (e.g., spinal fusion, metal implants, etc.), severe scoliosis and severe degenerative changes (e.g., osteophytes, sclerosis)
* Bilateral hip replacement
* Any restrictions, defined by site requirements for hrMRI procedure (for subset of hrMRI subjects)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (39):
- United States (39):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Gainsville, Georgia
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, South Portland, Maine
  - GSK Investigational Site, Bathesda, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Beckley, West Virginia
  - GSK Investigational Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo orally at a dose of 150 mg once a month for 12 months
- Ibandronate: Ibandronate orally at a dose of 150 mg once a month for 12 months
Period: Overall Study
Arm/Group | Placebo | Ibandronate
Started | 48 | 87
Completed | 41 | 69
Not Completed | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibandronate | Total
Number analyzed (Participants) | 47 | 85 | 132
Age, Customized [Number; unit: participants] — Safety analysis population
  participants
    < 65 years | 23 | 42 | 65
    >= 65 years | 24 | 43 | 67
Age Continuous [Mean (Standard Deviation); unit: years] — Safety analysis population
  years | 65.0 (10.63) | 63.9 (11.20) | 64.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety analysis population
  Participants
    Female | 0 | 0 | 0
    Male | 47 | 85 | 132

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in BMD of the Lumbar Spine From Baseline to Month 12
Description: BMD will be assessed using an analysis of covariance model (ANCOVA) with datea obtained from dual-Energy X-ray absorptiometry scans.
Time Frame: 12 months
Population: Intent-to-treat population. Includes participants with measurements at Baseline and Month 12.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Ibandronate
Number analyzed (Participants) | 42 | 77
percent | .94 (0.709) | 3.52 (0.661)
Statistical Analysis 1: Comparison: Placebo vs Ibandronate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 2.58, 95% CI [1.41 to 3.76]

2. Secondary Outcome: Mean Percent Change in BMD of the Lumbar Spine From Baseline to Month 6
Description: as for outcome 1
Time Frame: 6 months
Population: Intent-to-treat population. Includes patients with measurements at Baseline and Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Ibandronate
Number analyzed (Participants) | 41 | 77
percent | 0.78 (0.649) | 1.64 (0.604)
Statistical Analysis 1: Comparison: Placebo vs Ibandronate; Test type: Superiority or Other; p = 0.118, ANCOVA; Mean Difference (Net) = 0.86, 95% CI [-0.22 to 1.94]

3. Secondary Outcome: Mean Percent Change in BMD of Proximal Femur Sites (Total Hip, Trochanter, Femoral Neck) From Baseline to Month 12
Description: as for outcome 1
Time Frame: 12 months
Population: Intent-to-treat population. Includes patients with measurements at Baseline and Month 12.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Ibandronate
Number analyzed (Participants) | 42 | 77
percent
  Total Hip | -0.31 (0.473) | 1.82 (0.430)
  Femoral Neck | -0.23 (0.663) | 1.21 (0.612)
  Trochanter | 0.43 (0.692) | 2.15 (0.633)
Statistical Analysis 1: Comparison: Placebo vs Ibandronate; Total Hip subgroup; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 2.13, 95% CI [1.34 to 2.92]
Statistical Analysis 2: Comparison: Placebo vs Ibandronate; Femoral Neckm subgroup; Test type: Superiority or Other; p = 0.012, ANCOVA; Mean Difference (Net) = 1.43, 95% CI [0.32 to 2.55]
Statistical Analysis 3: Comparison: Placebo vs Ibandronate; Trochanter subgroup; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Net) = 1.72, 95% CI [0.56 to 2.88]

4. Secondary Outcome: Mean Percent Change in BMD of Proximal Femur Sites (Total Hip, Trochanter, Femoral Neck) From Baseline to Month 6
Description: as for outcome 1
Time Frame: 6 months
Population: Intent-to-treat population. Includes patients with measurements at Baseline and Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Ibandronate
Number analyzed (Participants) | 41 | 77
percent
  Total Hip | -0.48 (0.386) | 1.27 (0.349)
  Femoral Neck | -0.22 (0.630) | 0.96 (0.580)
  Trochanter | 0.55 (0.677) | 2.59 (0.616)
Statistical Analysis 1: Comparison: Placebo vs Ibandronate; Total Hip subgroup; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 1.75, 95% CI [1.11 to 2.40]
Statistical Analysis 2: Comparison: Placebo vs Ibandronate; Femoral Neck subgroup; Test type: Superiority or Other; p = 0.031, ANCOVA; Mean Difference (Net) = 1.18, 95% CI [0.11 to 2.25]
Statistical Analysis 3: Comparison: Placebo vs Ibandronate; Trochanter subgroup; Test type: Superiority or Other; p = 0.031, ANCOVA; Mean Difference (Net) = 1.18, 95% CI [0.11 to 2.25]

5. Secondary Outcome: Responder Rate of Subjects Who Remained the Same or Had Any Improvement in BMD (>= Baseline) at 6 Months and 12 Months
Description: Responders are defined as participants who have BMD values >= their baseline values at Months 6 and 12, and not any pre-defined percentage increase in BMD values of clinical significance.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: participants
Arm/Group | Placebo | Ibandronate
Number analyzed (Participants) | 47 | 85
participants
  Month 6: Lumbar Spine | 30 | 62
  Month 6: Total Hip | 14 | 57
  Month 6: Lumbar Spine and Total Hip | 10 | 46
  Month 12: Lumbar Spine | 33 | 71
  Month 12: Total Hip | 20 | 64
  Month 12: Lumbar Spine and Total Hip | 16 | 59
Statistical Analysis 1: Comparison: Placebo vs Ibandronate; Total Spine BMD at Month 6; Test type: Superiority or Other; p = 0.362, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.91, 95% CI [0.73 to 1.13] — Relative risk
Statistical Analysis 2: Comparison: Placebo vs Ibandronate; Total Spine BMD at Month 12; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.85, 95% CI [0.72 to 1.01] — Relative risk
Statistical Analysis 3: Comparison: Placebo vs Ibandronate; Total Hip BMD at Month 6; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.46, 95% CI [0.30 to 0.72] — Relative risk
Statistical Analysis 4: Comparison: Placebo vs Ibandronate; Total Hip BMD at Month 12; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.57, 95% CI [0.41 to 0.80] — Relative risk
Statistical Analysis 5: Comparison: Placebo vs Ibandronate; Both Total Hip and Total Spine BMD at Month 6; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.41, 95% CI [0.23 to 0.72] — Relative risk
Statistical Analysis 6: Comparison: Placebo vs Ibandronate; Both Total Hip and Total Spine BMD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.50, 95% CI [0.33 to 0.75] — Relative risk

ADVERSE EVENTS:
Description: Safety analysis population
Arm/Group | Placebo | Ibandronate
Serious Adverse Events (participants affected / at risk) | 6/47 | 7/86
Other Adverse Events (participants affected / at risk) | 13/47 | 27/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | Ibandronate (N=86)
Death (General disorders) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Multiple sclerosis (Nervous system disorders) | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Renal failure actue (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | Ibandronate (N=86)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 7
Constipation (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No